CLINICAL TRIAL: NCT05639127
Title: Novel Treatment of Adrenal Crisis: an Early Clinical Trial With Nebulized Prednisolone
Brief Title: The Treatment of Adrenal Crisis With Inhaled Prednisolone
Acronym: TRACER
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL81816.056.22
Record Dates: First submitted 2022-08-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-08

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: Open label single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low dose, wash out, high dose (Experimental)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Nebulization of prednisolone

SUMMARY:
Rationale: An adrenal crisis is an acute life-threatening event which may occur in patients with adrenal insufficiency. The initial emergency treatment consists of an intramuscular injection with 100 mg hydrocortisone administered by the patient or a bystander. The injection should be administered immediately. Although it is considered life-saving, it is not very patient-friendly, because of the several steps required for reconstitution, the intramuscular injection, the frequent presence of needle phobia, and pain at the injection site. Inhalation of predniso(lo)ne could be a more patient-friendly alternative.

Objective: This study investigates the pharmacokinetics of nebulized prednisolone in two different dosages.

Study design: Single-center, open-label study Study population: Healthy participants aged 18-75 years. Intervention (if applicable): Healthy volunteers receive a lower dose of nebulized prednisolone (46.75 mg).After a wash-out period of at least one week, each volunteer receives a higher dose of nebulized prednisolone (93.5 mg).

Main study parameters/endpoints: To establish the time from nebulizing to maximum prednisolone concentration in serum and the area under the curve of prednisolone.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants are exposed to a single supraphysiological dose of glucocorticoids on two separate occasions. The risk of SAE is very limited. There is a small risk of an AE during blood sampling. If it is demonstrated that therapeutic plasma concentrations of prednisolone can be reached by nebulizing prednisolone, we intend to use the pharmacokinetic data to design and perform a clinical study with a dry-powder micronized prednisone inhalation. This would represent a novel and promising alternative treatment for an adrenal crisis. Patients with adrenal insufficiency could then be offered a much more patient-friendly and reliable alternative for intramuscular hydrocortisone injection.

DETAILED DESCRIPTION:
The prevalence of adrenal insufficiency is approximately 30-50 individuals per 100.0001. Patients with adrenal insufficiency rely on glucocorticoid substitution therapy (hydrocortisone or cortisone acetate). In case of an acute stressful situation, e.g. illness, trauma, or psychological stress, the standard substitution dose falls short and patients need to increase their glucocorticoid dose to prevent a cortisol deficiency which could ultimately lead to an adrenal crisis. The incidence of an adrenal crisis is about 5-10 cases per year 100 patient-years and is characterized by hypotension, nausea, hyponatremia, hyperkalemia, hypoglycemia, and a circulatory shock with the risk of a fatal outcome2,3. Acute glucocorticoid administration in case of an adrenal crisis is a life-saving procedure.

Currently, patients have to inject themselves with an intramuscular injection of hydrocortisone sodium succinate, corresponding with 100 mg hydrocortisone. This mode of self-treatment has several disadvantages. Hydrocortisone sodium succinate is an unstable product in solution, it is therefore available as Solu-cortef Act-O-Vial in two-chamber vials containing hydrocortisone powder and diluent solution separately. The patient should first prepare the solution and then self-administer the hydrocortisone solution by an intramuscular injection. This is a multistep procedure (Supplement 1). If the injected dose is insufficient, a second injection might be necessary.

In addition, patients with an (imminent) adrenal crisis often experience confusion, drowsiness, dizziness, and nausea with vomiting. As a result, patients may be incapacitated to self-administer intramuscular hydrocortisone. Moreover, needle phobia might hamper self-injection of hydrocortisone. Furthermore, patients are advised to always carry the Solu-Cortef® Act-O-vial, syringe, and needles with them. This is, however, often not very practical and many patients do not follow up on this recommendation. These disadvantages of self-injection of hydrocortisone create a barrier for optimal emergency treatment. It is therefore logical that this method of drug administration is often not sufficiently used and easily leads to errors. Notably, we recently published data about adrenal crises in our own UMCG population and concluded that less than half of the patients who experienced an adrenal crisis used their emergency medication4.

A small inhalation device containing micronized prednisone seems a promising alternative for the replacement of the hydrocortisone injection. It is known that several drugs have a similar time from administration to effect after inhalation as after injection. Examples are adrenaline, levodopa, morphine, and insulin5. Based on its physicochemical properties, prednisone is expected to be as rapidly distributed into the bloodstream after inhalation compared to an intramuscular injection. In addition, previous application of inhaled prednisone for patients with asthma and COPD has demonstrated that the inhalation of prednisone is safe6.

A major advantage to prednisone inhalation compared to the Solu-Cortef® injection is that difficult reconstitution procedures are no longer necessary. In addition, the prednisone powder within the inhalator is very stable and easy to carry along as it fits inside a small pocket. Moreover, in contrast to intramuscular self-injection, inhalation treatment is pain-free and is expected to be acceptable for the majority of patients The patient's resistance against inhalation is much less than against the injection.

As the first step in the development of this prednisone inhaler we will investigate if therapeutic plasma concentrations of prednisolone can be reached by nebulizing prednisolone. In this study, we administer nebulized prednisolone in two different dosages to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years
* Woman who use reliable contraceptives or with a negative pregnancy test
* Equal sex distribution

Exclusion Criteria:

* Heart failure
* Known liver or kidney disease
* Dependency on glucocorticoids
* Adrenogenital syndrome
* Infectious disease
* Uncontrolled hypertension defined as a blood pressure > 180/110 mmHg
* Pregnancy or breastfeeding
* Use of medication that interferes with cytochrome P450 (e.g. carbamazepine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Tmax | 4 hours
  The time from nebulization to peak concentration prednisolone (Tmax (min))
AUC | 4 hours
  The area under the curve (AUC (h*nmol/L))

SECONDARY OUTCOMES:
Cmax | 4 hours
  Peak concentration (Cmax (nmol/L))
T1/2 | 4 hours
  Half life (T1/2 (h))
CL | 4 hours
  Total Body Clearance (CL (L/h))
Vd | 4 hours
  Volume of distribution (Vd (L))

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion study
Access Criteria: Upon reasonable request